CLINICAL TRIAL: NCT00783263
Title: A Multicenter, Randomized, Double-Blind, Titration Study to Evaluate the Efficacy and Safety of Ezetimibe Added On to Rosuvastatin Versus Up Titration of Rosuvastatin in Patients With Hypercholesterolemia at Risk for Coronary Heart Disease
Brief Title: A Study of Ezetimibe Added On to Rosuvastatin Versus Up Titration of Rosuvastatin in Patients With Hypercholesterolemia (MK0653-139)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-139; 2008_567
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2011-09-14 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rosuvastatin 5 mg + Ezetimibe 10 mg (Experimental): Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 5 mg rosuvastatin for an additional 6 weeks.
  Interventions: Drug: Comparator: rosuvastatin 5 mg + ezetimibe 10 mg
- Rosuvastatin 10 mg (Active Comparator): Participants who received rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 10 mg once daily for 6 additional weeks.
  Interventions: Drug: Comparator: rosuvastatin 10 mg
- Rosuvastatin 10 mg + Ezetimibe 10 mg (Experimental): Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 10 mg rosuvastatin for an additional 6 weeks.
  Interventions: Drug: Comparator: rosuvastatin 10 mg + ezetimibe 10 mg
- Rosuvastatin 20 mg (Active Comparator): Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 20 mg once daily for 6 additional weeks.
  Interventions: Drug: Comparator: rosuvastatin 20 mg

INTERVENTIONS:
Drug: Comparator: rosuvastatin 5 mg + ezetimibe 10 mg — Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 5 mg rosuvastatin for an additional 6 weeks.
  Other Names: Crestor, Zetia
  Arms: Rosuvastatin 5 mg + Ezetimibe 10 mg
Drug: Comparator: rosuvastatin 10 mg — Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 10 mg once daily for 6 additional weeks.
  Other Names: Crestor
  Arms: Rosuvastatin 10 mg
Drug: Comparator: rosuvastatin 10 mg + ezetimibe 10 mg — Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 10 mg rosuvastatin for an additional 6 weeks.
  Other Names: Crestor, Zetia
  Arms: Rosuvastatin 10 mg + Ezetimibe 10 mg
Drug: Comparator: rosuvastatin 20 mg — Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 20 mg once daily for 6 additional weeks.
  Other Names: Crestor
  Arms: Rosuvastatin 20 mg

SUMMARY:
A study to evaluate the low-density lipoprotein cholesterol (LDL-C) lowering efficacy of the addition of ezetimibe to rosuvastatin compared with doubling dose of rosuvastatin in participants treated with rosuvastatin alone and not at their National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) LDL-C goal

ELIGIBILITY:
Inclusion Criteria:

* Participant is currently taking a stable dose of lipid lowering agent(s). (if applicable) or is statin naive
* Participant is currently taking a stable dose of lipid lowering agent(s). (if is at least moderate high risk for Coronary Heart Disease (CHD))
* Participant is currently taking a stable dose of lipid lowering agent(s). (if is willing to maintain Therapeutic Lifestyle Changes (TLC) / American Diabetes Association(ADA) diet)

Exclusion Criteria:

* Participant weighs less than 100 lbs (45 kg).
* Participant has hypersensitivity or intolerance to ezetimibe, or rosuvastatin or any components of these medications.
* If female, participant is pregnant or breastfeeding.
* Participant consumes more than 2 alcoholic beverages per day.
* Participant has been in a clinical trial within the last 30 days.
* Participant has heart problems such as CHF, unstable angina or heart attack.
* Participant has type 1 or 2 diabetes and has changed their medication in the last 2 months.
* Participant has liver disease.
* Participant is Human Immunodeficiency Virus (HIV) positive.
* Participant has a history of drug or alcohol abuse in the last year.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bays HE, Davidson MH, Massaad R, Flaim D, Lowe RS, Tershakovec AM, Jones-Burton C. Safety and efficacy of ezetimibe added on to rosuvastatin 5 or 10 mg versus up-titration of rosuvastatin in patients with hypercholesterolemia (the ACTE Study). Am J Cardiol. 2011 Aug 15;108(4):523-30. doi: 10.1016/j.amjcard.2011.03.079. Epub 2011 May 17. PMID 21596364

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosuvastatin 10 mg: Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 10 mg once daily for 6 additional weeks.
Period: Overall Study
Arm/Group | Rosuvastatin 5 mg + Ezetimibe 10 mg | Rosuvastatin 10 mg | Rosuvastatin 10 mg + Ezetimibe 10 mg | Rosuvastatin 20 mg
Started | 99 | 98 | 122 | 121
Completed | 95 | 96 | 119 | 118
Not Completed | 4 | 2 | 3 | 3
Not completed — Adverse Event | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 5 mg + Ezetimibe 10 mg | Rosuvastatin 10 mg | Rosuvastatin 10 mg + Ezetimibe 10 mg | Rosuvastatin 20 mg | Total
Number analyzed (Participants) | 99 | 98 | 122 | 121 | 440
Age, Customized [Number; unit: participants]
  < 65 years | 63 | 62 | 71 | 71 | 267
  ≥ 65 years | 36 | 36 | 51 | 50 | 173
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 56 | 37 | 168
  Male | 64 | 58 | 66 | 84 | 272

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-Cholesterol (mg/dL) After 6 Weeks of Treatment
Description: The percent change from baseline in LDL-C (mg/dL) after 6 weeks of treatment in participants who were administered ezetimibe 10 mg to rosuvastatin (5 or 10 mg) in comparison with doubling the baseline dose of rosuvastatin (10 or 20 mg) daily for 6 weeks.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg: Participants who received open label rosuvastatin (5 or 10 mg) tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus (5 or 10 mg) rosuvastatin for an additional 6 weeks.
- Rosuvastatin (10 or 20 mg): Participants who received open label rosuvastatin (5 or 10 mg) tablets once daily for 4 to 5 weeks then received rosuvastatin (10 or 20 mg) once daily for 6 additional weeks.
Arm/Group | Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg | Rosuvastatin (10 or 20 mg)
Number analyzed (Participants) | 219 | 217
percent change | -21.57 (25.09) | -5.58 (25.42)
Statistical Analysis 1: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin (10 or 20 mg); Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis (LDA); Longitudinal Data Analysis was based on a constrained LDA model with terms for treatment, time, stratum and the interaction of time by treatment; Mean Difference (Final Values) = -15.25, 95% CI 2-sided [-19.89 to -10.60]

2. Secondary Outcome: Percent Change From Baseline in LDL-Cholesterol (mg/dL) After 6 Weeks of Treatment in Each Stratum
Description: The percent change from baseline in LDL-C (mg/dL) after 6 weeks of treatment by stratum I and stratum II in participants who were administered with ezetimibe 10 mg to rosuvastatin (5 or 10 mg) in comparison with the doubling of the baseline dose of rosuvastatin (10 or 20 mg) daily for 6 weeks.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Rosuvastatin 5 mg + Ezetimibe 10 mg (Stratum I): Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 5 mg rosuvastatin for an additional 6 weeks.
- Rosuvastatin 10 mg (Stratum I); Rosuvastatin 10 mg + Ezetimibe 10 mg (Stratum II): Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 10 mg once daily for 6 additional weeks.
- Rosuvastatin 20 mg (Stratum II): Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 20 mg once daily for 6 additional weeks.
Arm/Group | Rosuvastatin 5 mg + Ezetimibe 10 mg (Stratum I) | Rosuvastatin 10 mg (Stratum I) | Rosuvastatin 10 mg + Ezetimibe 10 mg (Stratum II) | Rosuvastatin 20 mg (Stratum II)
Number analyzed (Participants) | 98 | 96 | 121 | 121
percentage change | -18.57 (26.35) | -4.96 (22.42) | -24.00 (23.86) | -6.07 (27.65)
Statistical Analysis 1: Comparison: Rosuvastatin 5 mg + Ezetimibe 10 mg (Stratum I) vs Rosuvastatin 10 mg (Stratum I); Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis (LDA); Longitudinal Data Analysis was based on a constrained LDA model with terms for treatment, time and the interaction of time by treatment; Mean Difference (Final Values) = -12.31, 95% CI 2-sided [-18.95 to -5.67]
Statistical Analysis 2: Comparison: Rosuvastatin 10 mg + Ezetimibe 10 mg (Stratum II) vs Rosuvastatin 20 mg (Stratum II); Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis (LDA); [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -17.46, 95% CI 2-sided [-23.92 to -10.99]

3. Secondary Outcome: Number of Participants Who Reached Their Target LDL-C Level
Description: Participants were analyzed to evaluate the LDL-C (<100 mg/dL for moderately high risk patients and high risk patients without AVD and <70 mg/dL for high risk patients with AVD) lowering efficacy with the addition of ezetimibe 10 mg to (5 or 10 mg) compared with doubling the baseline rosuvastatin (10 or 20 mg), daily for 6 weeks of treatment.
Time Frame: 6 weeks of treatment
Measure: Number; unit: participants
Groups:
- Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg: Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 5 mg rosuvastatin for an additional 6 weeks.
- Rosuvastatin (10 or 20 mg): Participants who received rosuvastatin (5 or 10 mg) mg tablets once daily for 4 to 5 weeks then received rosuvastatin (10 or 20 mg) once daily for 6 additional weeks.
Arm/Group | Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg | Rosuvastatin (10 or 20 mg)
Number analyzed (Participants) | 219 | 217
participants | 130 | 67
Statistical Analysis 1: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin (10 or 20 mg); Test type: Superiority or Other; p < 0.001, Logistic Regression; Logistic Regression included terms for treatment, stratum and baseline LDL-C category (3 levels: <100, 100-<130, ≥130 mg/dL); Odds Ratio (OR) = 4.5, 95% CI 2-sided [2.9 to 6.9]

4. Secondary Outcome: Number of Participants in Each Stratum Who Reached Their Target LDL-C Level
Description: Participants in stratum I were analyzed to evaluate the LDL-C lowering efficacy with the additional of ezetimibe 10 mg to rosuvastatin 5 mg daily for 6 weeks compared with doubling the baseline dose to rosuvastatin 10 mg daily for 6 weeks. Participants in stratum II were analyzed to evaluate the LDL-C lowering efficacy with the additional of ezetimibe 10 mg to rosuvastatin 10 mg daily for 6 weeks compared with doubling the baseline dose to rosuvastatin 20 mg daily for 6 weeks.
Time Frame: 6 weeks of treatment
Measure: Number; unit: participants
Groups:
- Rosuvastatin 5 mg + Ezetimibe 10 mg (Stratum I); Rosuvastatin 10 mg + Ezetimibe 10 mg (Stratum II): Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 10 mg rosuvastatin for an additional 6 weeks.
- Rosuvastatin 10 mg (Stratum I); Rosuvastatin 20 mg (Stratum II): Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 20 mg once daily for 6 additional weeks.
Arm/Group | Rosuvastatin 5 mg + Ezetimibe 10 mg (Stratum I) | Rosuvastatin 10 mg (Stratum I) | Rosuvastatin 10 mg + Ezetimibe 10 mg (Stratum II) | Rosuvastatin 20 mg (Stratum II)
Number analyzed (Participants) | 98 | 96 | 121 | 121
participants | 54 | 30 | 76 | 37
Statistical Analysis 1: Comparison: Rosuvastatin 5 mg + Ezetimibe 10 mg (Stratum I) vs Rosuvastatin 10 mg (Stratum I); Test type: Superiority or Other; p < 0.001, Logistic Regression; Logistic Regression included terms for treatment and baseline LDL-C category (3 levels: <100, 100-<130, >=130 mg/dL); Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.7 to 5.8]
Statistical Analysis 2: Comparison: Rosuvastatin 10 mg + Ezetimibe 10 mg (Stratum II) vs Rosuvastatin 20 mg (Stratum II); Test type: Superiority or Other; p < 0.001, Logistic Regression; Logistic Regression included terms for treatment and baseline LDL-C category (3 levels: <100, 100-<130, >=130 mg/dL); Odds Ratio (OR) = 6.5, 95% CI 2-sided [3.4 to 12.3]

5. Secondary Outcome: Number of Participants Who Reached the LDL-C Level of <70 mg/dl
Description: Participants across all strata who reached the LDL-C Level of <70 mg/dl after the addition of ezetimibe 10 mg to rosuvastatin (5 or 10 mg) daily for 6 weeks compared with doubling the baseline dose of rosuvastatin (10 or 20 mg) daily for 6 weeks.
Time Frame: 6 weeks of treatment
Measure: Number; unit: participants
Groups:
- Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg: Participants who received open label rosuvastatin 5 or 10 mg tablets once daily for 4 to 5 weeks then received 10 or 20 mg ezetimibe tablets once daily plus 5 mg rosuvastatin for an additional 6 weeks.
- Rosuvastatin 10 or 20 mg: Participants who received rosuvastatin (5 or 10 mg) tablets once daily for 4 to 5 weeks then received rosuvastatin (10 or 20 mg) once daily for 6 additional weeks.
Arm/Group | Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg | Rosuvastatin 10 or 20 mg
Number analyzed (Participants) | 219 | 217
participants | 96 | 38
Statistical Analysis 1: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression; Odds Ratio (OR) = 8.0, 95% CI 2-sided [4.6 to 14.0]

6. Secondary Outcome: Number of Participants in Each Stratum Who Reached the LDL-C Level of <70 mg/dl
Description: Participants in stratum I and in stratum II who reached the LDL-C Level of <70 mg/dl after the addition of ezetimibe to rosuvastatin (5 or 10 mg)daily for 6 weeks compared with doubling the baseline dose of rosuvastatin (10 or 20 mg).
Time Frame: 6 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Rosuvastatin 5 mg + Ezetimibe 10 mg | Rosuvastatin 10 mg | Rosuvastatin 10 mg + Ezetimibe 10 mg | Rosuvastatin 20 mg
Number analyzed (Participants) | 98 | 96 | 121 | 121
participants | 31 | 12 | 65 | 26
Statistical Analysis 1: Comparison: Rosuvastatin 5 mg + Ezetimibe 10 mg vs Rosuvastatin 10 mg; Stratum I; Test type: Superiority or Other; p < 0.001, Logistic Regression; Odds Ratio (OR) = 5.1, 95% CI 2-sided [2.2 to 11.8]
Statistical Analysis 2: Comparison: Rosuvastatin 10 mg + Ezetimibe 10 mg vs Rosuvastatin 20 mg; Stratum II; Test type: Superiority or Other; p < 0.001, Logistic Regression; Odds Ratio (OR) = 11.4, 95% CI 2-sided [5.2 to 24.8]

7. Secondary Outcome: Percent Change From Baseline in Other Lipid, Lipoprotein, Apolipoprotein and High-sensitivity C-reactive Protein (Hs-CRP)Levels
Description: Participants who were analyzed to assess the Total Cholesterol (TC), Triglycerides, High-Density Lipoprotein Cholesterol, Non High-Density Lipoprotein Cholesterol, LDL Cholesterol/HDL Cholesterol, Total Cholesterol/HDL Cholesterol, Non-HDL Cholesterol/HDL Cholesterol, Apolipoprotein B (Apo B), Apolipoprotein A-I (Apo A-I), Apolipoprotein B/Apo A-I, high-sensitivity C-reactive protein (hs-CRP)levels after 6 weeks of treatment.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg | Rosuvastatin 10 or 20 mg
Number analyzed (Participants) | 219 | 217
percentage change
  Total Cholesterol (TC) | -13.00 (17.51) | -3.76 (14.35)
  Triglycerides | -5.96 (36.45) | -3.60 (32.83)
  High-Density Lipoprotein Cholesterol | -0.67 (15.51) | 2.18 (13.38)
  Non High-Density Liproprotein Cholesterol | -17.59 (23.55) | -5.29 (21.20)
  LDL Cholesterol/HDL Cholesterol | -19.48 (27.63) | -6.18 (27.82)
  Total Cholesterol/HDL Cholesterol | -10.57 (25.87) | -4.40 (18.27)
  Non-HDL Cholestrol/HDL Cholesterol | -14.51 (35.39) | -5.31 (26.63)
  Apolipoprotein B (Apo B) | -14.31 (18.61) | -4.25 (17.56)
  Apolipoprotein A-I (Apo A-I) | -1.44 (12.49) | 1.06 (11.56)
  Apolipoprotein B/Apo A-I | -11.98 (20.84) | -4.11 (19.61)
  hs-C-Reactive Protein | -13.98 (72.19) | -12.82 (73.08)
Statistical Analysis 1: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Total Cholesterol (mg/dL); Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -8.65, 95% CI 2-sided [-11.59 to -5.71]
Statistical Analysis 2: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Triglycerides (mg/dL); Test type: Superiority or Other; p = 0.306, Longitudinal Data Analysis; Mean Difference (Final Values) = -3.10, 95% CI 2-sided [-9.04 to 2.84]
Statistical Analysis 3: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; High-Density Lipoprotein Cholesterol; Test type: Superiority or Other; p = 0.111, Longitudinal Data Analysis; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-4.79 to 0.49]
Statistical Analysis 4: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Non High-Density Liproprotein Cholesterol; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -11.98, 95% CI 2-sided [-16.10 to -7.86]
Statistical Analysis 5: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; LDL Cholesterol/HDL Cholesterol; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -13.25, 95% CI 2-sided [-18.36 to -8.13]
Statistical Analysis 6: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Total Cholesterol/HDL Cholesterol; Test type: Superiority or Other; p = 0.002, Longitudinal Data Analysis; Mean Difference (Final Values) = -6.45, 95% CI 2-sided [-10.53 to -2.36]
Statistical Analysis 7: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Non-HDL Cholestrol/HDL Cholesterol; Test type: Superiority or Other; p = 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -9.52, 95% CI 2-sided [-15.30 to -3.75]
Statistical Analysis 8: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Apolipoprotein B (Apo B); Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -9.41, 95% CI 2-sided [-12.74 to -6.08]
Statistical Analysis 9: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Apolipoprotein A-I (Apo A-I); Test type: Superiority or Other; p = 0.102, Longitudinal Data Analysis; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-3.99 to 0.36]
Statistical Analysis 10: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; Apolipoprotein B/Apo A-I; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -7.54, 95% CI 2-sided [-11.25 to -3.83]
Statistical Analysis 11: Comparison: Rosuvastatin (5 or 10 mg) + Ezetimibe 10 mg vs Rosuvastatin 10 or 20 mg; hs-C-Reactive Protein; Test type: Superiority or Other; p = 0.861, Longitudinal Data Analysis; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-13.13 to 10.97]

ADVERSE EVENTS:
Description: All participants randomized were treated and had safety follow up.
Groups:
- Rosuva 5 mg + EZ 10 mg: Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 5mg rosuvastatin for an additional 6 weeks.
- Rosuva 10 mg: Participants who received open label rosuvastatin 5 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 10 mg once daily for 6 additional weeks.
- Rosuva 10 mg + EZ 10 mg: Participants who received open label rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received 10 mg ezetimibe tablets once daily plus 10 mg rosuvastatin for an additional 6 weeks.
- Rosuva 20 mg: Participants who received rosuvastatin 10 mg tablets once daily for 4 to 5 weeks then received rosuvastatin 20 mg once daily for 6 additional weeks.
Arm/Group | Rosuva 5 mg + EZ 10 mg | Rosuva 10 mg | Rosuva 10 mg + EZ 10 mg | Rosuva 20 mg
Serious Adverse Events (participants affected / at risk) | 0/99 | 1/98 | 0/122 | 1/121
Other Adverse Events (participants affected / at risk) | 0/99 | 0/98 | 0/122 | 0/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuva 5 mg + EZ 10 mg (N=99) | Rosuva 10 mg (N=98) | Rosuva 10 mg + EZ 10 mg (N=122) | Rosuva 20 mg (N=121)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less